CLINICAL TRIAL: NCT06147206
Title: "ANTES" Proposal: A New Approach to Exacerbation in COPD Patients. Exacerbantes Study.
Brief Title: Exacerbantes Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Juan José Soler Cataluna, MD, Pneumologist, Sociedad Española de Neumología y Cirugía Torácica
Other Study IDs: NEM_EPOC_2023.1
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: COPD Exacerbation
Keywords: COPD; Exacerbation; Personalized medicine; Treatable traits
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample to assess several biomarkers (CRP, NT-proBNP, Troponin) in hospital emergence treated population. Only capillary CRP in the primary care treated population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) is understood as a complex and heterogeneous syndrome, which requires an increasingly personalized approach. A new approach to AECOPD recognized that several etiopathogenic mechanisms can lead to a worsening ot the patients. This new approach is based on the identification of different treatable traits (TTs).

The goal of this observational study is to describe how TTs are distributed in patients with AECOPD in primary care (PC) and hospital emergencies department (HED) to address their complexity and heterogeneity.

As a secondary outcomes we also try to evaluate the relationship of TTs with relevant clinical outcomes (relapse, recurrence, MACE (Major Adverse Cardiovascular Event) and all-cause mortality) and create a risk score and compare this new severity score with Rome and GesEPOC proposals.

In the AP group, a series of basic tests for routine use will be systematically performed, among which chest x-ray, electrocardiogram and other new tests such as microspirometry (COPD-6) and a point of care determination of capillary C-reactive protein (CRP). In the HED group routine determinations will be expanded to include blood tests, arterial blood gases and biomarkers (CRP, TnT, NT-proBNP and D-Dimer). Patients will be re-evaluated 90 days after the initial episode, to evaluate different clinical outcomes. The estimated sample size is 400 patients.

DETAILED DESCRIPTION:
Justification COPD exacerbations (AECOPD) are heterogeneous and complex in nature, demanding an increasingly personalized approach. Recently, the ANTES proposal was presented, a patient-centered approach based on the treatable traits (TT) strategy. Other recent initiatives, such as the Rome proposal or GesEPOC, also propose new definitions and ways to classify the severity of AECOPD. However, none of these 3 new proposals have been validated.

Objectives:

* Main: Describe in a systematic way how the different TTs are distributed in patients with AECOPD in primary care (PC) and hospital emergencies department (HED).
* Secondary: (1) evaluate the relationship of the different treatable features with the following clinical outcomes: relapse, recurrence, MACE (Major Adverse Cardiovascular Event) and all-cause mortality; (2) create a risk scale for recurrence, readmission, MACE and/or mortality, both in PC and HED; (3) compare the predictive capacity of the risk scale generated from the ANTES proposal, with the Rome and GesEPOC severity scales; (4): in the subgroup of patients treated in the hospital, compare the 3 risk scales (ANTES, Roma and GesEPOC) with the valid DECAF scale (5); assess whether it is feasible to determine FEV1, through the use of microspirometers, during COPD decompensation; and (6) compare lung function evaluated during decompensation with that obtained after recovery, 90 days after the index event.

Material:

Prospective, multicenter, longitudinal, observational study on patients diagnosed with AECOPD in PC and HED. In the AP cohort, a series of basic tests for routine use will be systematically performed, among which chest x-ray, electrocardiogram and other new tests such as microspirometry (COPD-6) and determination of point of care capillary C-reactive protein (CRP). In the HED cohort, routine determinations will be expanded to include blood tests, arterial blood gases and biomarkers (CRP, TnT, NT-proBNP and D-Dimer). Patients will be re-evaluated 90 days after the initial episode, to evaluate different clinical outcomes (relapse, recurrence, MACE and mortality). The distribution of different TTs will be analyzed and a new predictive risk scale will be created from them, comparing it with the Rome and GesEPOC scales. The estimated sample size is 400 patients.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who request emergency care (primary care or hospital) due to acute worsening of respiratory symptoms (of any nature)
* Age 40 years or older.
* Smokers or ex-smokers of > 10 pack-years
* Expiratory airflow limitation, documented by any of the following methods:

  * Post bronchodilation FEV1/FVC < 0.7, in a previous forced spirometry, or
  * FEV1/FEV6 less than 0.73 on microspirometry performed during decompensation

Exclusion Criteria:

* Patients with active neoplasia in the last 3 years.
* Associated pleural effusion susceptible to thoracentesis.
* Pneumothorax.
* Thoracic trauma.
* Impossibility of subsequent follow-up (3 months).

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COPD patients managed for worsening respiratory symptoms of any origin, both in primary care (PC group) and in the hospital emergency department (HED group) will be included.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
To describe treatable traits (TTs) distribution in AECOPD | Acute presentation of clinical worsening (less than 14 days)
  A treatable trait is defined as a clinical, functional or biological features, which can be identified through the use of diagnostic tests or biomarkers, and which have a specific treatment

SECONDARY OUTCOMES:
To evaluate the relationship of the different RTs with the following outcomes: relapse, recurrence, major adverse cardiovascular event (MACE) and mortality | 90 days of follow-up
  Relapse: appearance of a new worsening of symptoms within less than 4 weeks after the end of treatment for the index exacerbation; Recurrence: appearance of new worsening of symptoms beyond 4 weeks (during the 90 days of follow-up) after the end of treatment for the index exacerbation; • MACE (Major adverse cardiovascular event). The presence of at least one of the follow cardiovascular events in the 90 days after exacerbation index: acute myocardial infarct, unstable angor, revascularization, heart failure, stroke or cardiovascular mortality; Mortality: all-cause mortality in the 90 days of follow-up
To explore the creation of a predictive risk score (recurrence/ readmission/mortality/MACE) based on the patient-focused approach from the ANTES proposal in both PC and hospital emergency settings. | 90 days
  Risk score of severity
To compare the predictive capacity of the risk score generated from the ANTES proposal, with the Rome and GesEPOC severity scores | 90 days
  Rome and GesEPOC has a severity classification that will be compared with the new risk score created from ANTES proposal
In the subgroup of patients seen in hospital, compare the 3 risk score proposals (ANTES, Roma and GesEPOC) with the DECAF score | 90 days
  All 3 severity classifications will be compared with DECAF validated score, but only in those patients treated at hospital emergency room.
To assess the feasibility of FEV1 measurement by using a micro spirometer during COPD decompensation | During the first attendance of AECOPD (hours)
  Evaluate if FEV1 can be assessed during the AECOPD using COPD-6 microspirometer
6. To compare the lung function evaluated during COPD decompensation with that obtained after recovery, 90 days after the index event | 90 days
  Compared FEV1 values during AECOPD and stable phase 90 days after

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Soler-Cataluña, MD, Principal Investigator — Hospital Arnau de Vilanova (Valencia); Valencia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Celli BR, Fabbri LM, Aaron SD, Agusti A, Brook R, Criner GJ, Franssen FME, Humbert M, Hurst JR, O'Donnell D, Pantoni L, Papi A, Rodriguez-Roisin R, Sethi S, Torres A, Vogelmeier CF, Wedzicha JA. An Updated Definition and Severity Classification of Chronic Obstructive Pulmonary Disease Exacerbations: The Rome Proposal. Am J Respir Crit Care Med. 2021 Dec 1;204(11):1251-1258. doi: 10.1164/rccm.202108-1819PP. No abstract available. PMID 34570991
- [Background] Soler-Cataluna JJ, Pinera P, Trigueros JA, Calle M, Casanova C, Cosio BG, Lopez-Campos JL, Molina J, Almagro P, Gomez JT, Riesco JA, Simonet P, Rigau D, Soriano JB, Ancochea J, Miravitlles M; en representacion del grupo de trabajo de GesEPOC 2021. Spanish COPD Guidelines (GesEPOC) 2021 Update Diagnosis and Treatment of COPD Exacerbation Syndrome. Arch Bronconeumol. 2022 Feb;58(2):159-170. doi: 10.1016/j.arbres.2021.05.011. Epub 2021 May 26. English, Spanish. PMID 34172340
- [Background] Jose Soler-Cataluna J, Miravitlles M, Fernandez-Villar A, Izquierdo JL, Garcia-Rivero JL, Cosio BG, Lopez-Campos JL, Agusti A; ANTES panellists. Exacerbations in COPD: a personalised approach to care. Lancet Respir Med. 2023 Mar;11(3):224-226. doi: 10.1016/S2213-2600(22)00533-1. Epub 2023 Feb 10. No abstract available. PMID 36780913
- [Background] Soler-Cataluna JJ, Miralles C. Exacerbation Syndrome in COPD: A Paradigm Shift. Arch Bronconeumol (Engl Ed). 2021 Apr;57(4):246-248. doi: 10.1016/j.arbres.2020.07.008. Epub 2020 Sep 4. No abstract available. English, Spanish. PMID 32893033